CLINICAL TRIAL: NCT01513642
Title: Inspiratory Volume and Muscle Recruitment During Breath-stacking and Incentive Spirometry Techniques in Postoperative Cardiac Patients
Brief Title: Respiratory Physiotherapy After Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Juliana Flávia de Oliveira, Inspiratory Volume and Muscle Recruitment During Breath-stacking and Incentive Spirometry Techniques in Postoperative Cardiac Patients., Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: oliveira1
Record Dates: First submitted 2012-01-16; First posted 2012-01-20 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Functional Disturbance Following Cardiac Surgery
Keywords: physiotherapy; cardiac surgery; breath Stacking
MeSH Terms: interventions — Breathing Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Incentive spirometry (Other)
  Interventions: Behavioral: Breath Stacking
- Breath Stacking (No Intervention)

INTERVENTIONS:
Behavioral: Breath Stacking — To perform the BS maneuver, a silicone mask containing a one-way valve was attached to the patient's face. Once the mask was adjusted to allow only inspiration (the expiratory branch remained occluded), the patient was asked to make successive inspiratory efforts during 20 seconds.
  Other Names: respiratory exercises
  Arms: Incentive spirometry

SUMMARY:
Although incentive spirometry is commonly used to avoid pulmonary complications in cardiac surgery patients, the breath-stacking technique has been proposed as an alternative to increase pulmonary volumes in the post-operative period.

Objective: To compare inspiratory volume and electromyographic activity of respiratory muscles during breath stacking technique and incentive spirometry in patients undergoing cardiac surgery.

DETAILED DESCRIPTION:
The purpose of the present study are:

1. to evaluate and compare the inspiratory volume during the course of Breath Stacking and Incentive Spirometry techniques in patients submitted to myocardial revascularization surgery.
2. to compare the electromyographic activity of the scalene, sternocleidomastoid (SCM) and diaphragm muscles during both techniques.

ELIGIBILITY:
Inclusion Criteria:

* patients submitted to myocardial revascularization surgery

Exclusion Criteria:

* cognitive impairment or incoordination to perform IS
* face mask intolerance during BS
* level of consciousness incompatible to perform IS
* hemodynamic complications [arrhythmia, intraoperative myocardial infarction, major blood loss (defined as a loss of ≥20% of total blood volume), mean arterial pressure <70 mmHg and reduce cardiac output requiring the use of an intra-aortic balloon pump or vasoactive drugs)
* intubation for more than 72 h after admission to the Intensive Care Unit
* the need for reintubation.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-03; Primary Completion 2010-02 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Inspiratory volume and muscle recruitment during breath-stacking and incentive spirometry techniques in postoperative cardiac patients | Within 2 days after cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Dias, PhD, Study Director — Centro Universitário Augusto Motta
Locations (1):
- Federal Bonsucesso Hospital, Rio de Janeiro, Rio de Janeiro, Brazil